CLINICAL TRIAL: NCT01737645
Title: A Comparison of Intraocular Pressures (IOP) During Prolonged Trendelenburg Positioning in Morbidly Obese and Thin Patients
Status: Terminated | Type: Observational
Why Stopped: Difficulty in enrolling subjects.
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Roy Soto, MD, Principal Investigator, Corewell Health East
Other Study IDs: 2011-273
Record Dates: First submitted 2012-03-16; First posted 2012-11-29 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Intraocular Pressure Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- obese patients: BMI (body mass index) more than or equal to 35 kg/m2 (weight in kilograms divided by the square of the height in metres)
- Thin patients: BMI less than or equal to 30 kg/m2

SUMMARY:
This study is to determine if there is a rise in eye pressure, when patients are placed in a position where the head is lower than the rest of the body during long surgeries.

DETAILED DESCRIPTION:
Eye pressure will be measured at protocol specified intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing prolonged procedures (scheduled >3hr) in steep Trendelenburg position (eg. robotic prostatectomy, hysterectomy, cystectomy)
2. Morbidly obese subjects: BMI ≥ 35 kg/m2
3. Thin subjects: BMI ≤ 30 kg/m2
4. Age 18-70
5. ASA (American Society of Anesthesiologists) physical status classification I, II, or III

Exclusion Criteria:

1. Known history of glaucoma
2. Note:if initial IOP is noted to be >21mmHg (millimeters of mercury), patient will be excluded from study and an ophthalmology consultation will be obtained.Surgery will not be postponed.
3. Recent use of IOP lowering topical ophthalmic agents
4. Allergy to latex or proparacaine hydrochloride ophthalmic solution
5. Patients with active corneal epithelial defects or history of recurrent corneal erosion
6. Patients with underlying disorders that can directly increase intraocular pressure (thyroid eye disease, intra orbital tumors, orbital vascular malformation, Sturge-Weber disease, carotid or dural cavernous arteriovenous malformation, cavernous sinus pathology)
7. History of corneal surgery, to include LASIK (laser-assisted in-situ keratomileusis)
8. Any eye surgery within prior 1 month
9. Known pregnancy
10. Cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Subjects undergoing prolonged procedures expected to be in steep Trendelenburg position. Procedure must be scheduled for > 3 hours, eg. robotic prostatectomy, hysterectomy, and cystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To compare the percent change from baseline IOP reading to the peak IOP reading during steep Trendelenburg positioning in thin subjects vs morbidly obese subjects. | Measured from baseline IOP to peak IOP during steep Trendelenburg. The overall time frame for which the outcome measure is assessed is up to 3 years.

SECONDARY OUTCOMES:
To determine rate of rise of IOP during steep Trendelenburg positioning | The time during the surgery when the patient is in steep Trendelenburg positioning. The overall time frame for which the outcome measure is assessed is up to 3 years.
To compare peak IOP and rise of IOP during steep Trendelenburg positioning in thin vs morbidly obese subjects. | The time during the surgery when the patient is in steep Trendelenburg positioning. The overall time frame for which the outcome measure is assessed is up to 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Roy G Soto, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States